CLINICAL TRIAL: NCT03489629
Title: STaph Aureus Resistance-Treat Early and Repeat (STAR-TER)
Acronym: STAR-TER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Washington (Other); Cook Children's Medical Center (Other); Indiana University (Other); University of Michigan (Other); University of Texas Southwestern Medical Center (Other); St. Louis Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-2144
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cystic Fibrosis
Keywords: Methicillin-resistant Staphylococcus aureus (MRSA); Early infection; Treatment; Forced Expiratory Volume in 1 Second (FEV1)
MeSH Terms: conditions — Cystic Fibrosis; Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Minocycline; Mupirocin; chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Subjects are treated with one oral antibiotic, one topical antibiotic, an oral rinse, and instructed to use environmental decontamination techniques.
  Trimethoprim Sulfamethoxazole (TMP/SMX) is the primary oral antibiotic to be used. Subjects with allergy or intolerance to TMP_SMX will use minocycline as an alternative antibiotic. Topical antibiotics are nasal Mupirocin, and the oral rinse/gurgle with 0.12% chlorhexidine gluconate.
  Interventions: Drug: Trimethoprim Sulfamethoxazole (TMP/SMX); Drug: Minocycline; Drug: Mupirocin; Drug: Chlorhexidine Gluconate; Behavioral: Environmental Decontamination

INTERVENTIONS:
Drug: Trimethoprim Sulfamethoxazole (TMP/SMX) — Dosing if < 40 kg: 8 mg/kg trimethoprim/40 mg/kg trimethoprim sulfamethoxazole given twice daily for 14 days during Days 1-14 and Days 29-42.
  Dosing is ≥ 40 kg: 320 mg/1600 mg twice daily for 14 days during Days 1-14 and Days 29-42.
  Other Names: Septra; Bactrim
Drug: Minocycline — If a subject has an allergy to or intolerance to TMP/SMX, they may be treated with minocycline provided they are 8 years of age or older.
  Dosing if < 50 kg: 2 mg/kg orally twice daily for 14 days during Days 1-14 and Days 29-42.
  Dosing if ≥ 50 kg: 100 mg twice daily for 14 days during Days 1-14 and Days 29-42.
  Other Names: Cleeravue-M; Dynacin; Minocin; Solodyn; Vectrin
Drug: Mupirocin — 1 gram 2% nasal ointment generously applied to each nostril using a cotton swab twice daily for 5 days during Days 1-5 and Days 29-33.
  Other Names: Bactroban; Centany
Drug: Chlorhexidine Gluconate — For subjects able to swish without swallowing, 0.12% chlorhexidine gluconate oral rinse will be used twice daily for 14 days during Days 1-14 and Days 29-42.
  Other Names: Dyna-Hex
Behavioral: Environmental Decontamination — Subjects will be instructed to wipe down all high touch surfaces and medical equipment with surface disinfection wipes daily during Days 1-21 and Days 29-49.
  Subjects will also be instructed to wash all linens and towels in hot water once weekly during weeks 1-3 and weeks 5-7.
  Other Names: Sani-Cloth wipes

SUMMARY:
To evaluate the micro-biologic efficacy and safety of a streamlined treatment for early onset methicillin-resistant staphylococcus aureus (MRSA) in patients with cystic fibrosis.

DETAILED DESCRIPTION:
This is an open-label, multi-center interventional trial in Cystic Fibrosis (CF) patients with new MRSA isolated from the respiratory tract (oropharyngeal (OP) = OP swab, sputum, or bronchoscopy) at a clinical encounter.

Forty-two subjects with new MRSA infection will be enrolled and will receive two weeks of oral trimethoprim-sulfamethoxazole (TMP-SMX) or minocycline depending on age, allergies and antibiotic resistance of prior isolate for 14 days, and nasal mupirocin for 5 days. Subjects old enough to do so will use oral disinfectant gurgle (0.12% chlorhexidine gluconate oral rinse) for 14 days. The primary endpoint will be the proportion of positive MRSA respiratory cultures at Day 28 and this will be compared to our prior STAR-Too results.

Subjects will then have a 14 day wash-out period (i.e., no TMP-SMX or minocycline from Day 14 to Day 28) and all participants will repeat the treatment protocol from Day 29 to Day 42. Repeat cultures will be done at day 56 ± 7 days, most likely combined with their next clinic visit. Results of Day 56 cultures will be an exploratory, secondary outcome.

A subsequent visit will be 3 months later with their routine clinic appointment. Any interim clinic visits will be used to obtain repeat cultures and clinical data.

Assessment of MRSA culture status will be by OP swab for all subjects, with additional sputum in those who expectorate.

Total duration of an individual subject's participation will be six months. Total duration of the study is expected to be 42 months, which includes data analyses and publication.

Due to COVID 19 restrictions, a study amendment was filed in March 2020 for subjects currently active subjects that allowed remote study visit for V3 and V4. Cultures were collected at home and mailed to the Core Study lab, clinical case forms and surveys were completed via video visits. These changes were approved by each study site that this was relevant to i.e. 4 study sites had subjects active at that time.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 2 and ≤ 45 years of age at the Screening Visit.
2. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   1. sweat chloride ≥ 60 milliequivalents/liter by quantitative pilocarpine iontophoresis test (QPIT)
   2. two well-characterized mutations in the cystic fibrosis transmembrane conductive regulator (CFTR) gene
   3. abnormal nasal potential difference(NPD) (change in NPD in response to a low chloride solution and isoproteronol of less than -5 mV)
3. First OR early MRSA colonization defined as:

   1. First MRSA colonization: first documented isolation of MRSA from respiratory tract occurred ≤ 6 months prior to screening
   2. Early MRSA colonization: MRSA was previously isolated from the respiratory tract ≤ 2 times over the past 3.5 years, but this was followed by at least 1 year of documented negative cultures for MRSA
4. MRSA is available to the central laboratory - either the incident MRSA isolate from the clinic visit or the subject is MRSA positive at the screening visit
5. Clinically stable with no significant changes in health status within the 14 days prior to screening
6. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

1. Received antibiotics with activity against MRSA within 28 days prior to screening
2. Use of an investigational agent within 28 days prior to screening
3. For subjects ≥ 6 years of age: FEV1 at screening < 25% of predicted for age based on the Wang (males < 18 years, females < 16 years) or Hankinson (males ≥ 18 years, females ≥ 16 years) standardized equations
4. MRSA from the screening culture or the most recent clinical care visit within 6 months prior to screening resistant to TMP/SMX
5. History of intolerance to topical chlorhexidine or mupirocin
6. History of intolerance to both TMP/SMX and minocycline
7. < 8 years of age and allergic or intolerant to TMP/SMX
8. ≥ 8 years of age and allergic or intolerant to TMP/SMX and MRSA isolate (from screening or clinical care visit)is resistant to minocycline
9. For females of child bearing potential: pregnant, breastfeeding, or unwilling to use barrier contraception through Day 42 of the study
10. Subjects with history of abnormal renal function will need screening labs showing normal function Abnormal renal function is defined as estimated creatinine clearance <50 mL/min using the:

    1. Bedside Schwartz Equation for subjects <18 years of age, and
    2. Levey Glomerular filtration rate (GFR) Equation for subjects ≥ 18 years of age.
11. Subjects with a history of abnormal liver function will need to have screening labs showing normal transaminases. Liver dysfunction is defined as ≥3x upper limit of normal (ULN), of serum aspartate transaminase (AST) or serum alanine transaminase (ALT) or abnormal synthetic function
12. History of solid organ or hematological transplantation
13. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of STAR-TER subjects with a negative MRSA culture at Day 28 vs. observational arm of historic STAR-Too trial | Day 28
  Descriptive summary with corresponding 95% confidence interval.

SECONDARY OUTCOMES:
Proportion of subjects with a protocol-defined pulmonary exacerbation between Baseline and Day 28 treated with antibiotics active against MRSA | Period ranging from start of Baseline and continuing through Day 28
  Pulmonary exacerbation is defined as having 1 of the major criteria or 2 minor signs/symptoms and fulfillment of symptom duration.
  Major criteria:
  1. Absolute decrease in FEV1 of ≥ 10% from Visit 1 (Baseline), unresponsive to albuterol (in participants able to reproducibly perform spirometry)
  2. Oxygen saturation <90% on room air or absolute decrease of ≥ 5% from Visit 1
  3. New lobar infiltrate(s) or atelectasis on chest radiograph
  4. Hemoptysis (more than streaks on more than one occasion in past week)
  Minor signs/symptoms:
  1. Increased work of breathing or respiratory rate
  2. New or increased adventitial sounds on lung exam
  3. Weight loss ≥5% of body weight or decrease across 1 major percentile in weight percentile for age in past 6 months
  4. Increased cough
  5. Decreased exercise tolerance or level of activity
  6. Increased chest congestion or change in sputum
  Signs/symptoms duration: initial symptom must have occurred for at least 5 days.
Proportion of subjects with a protocol-defined pulmonary exacerbation between Baseline and Day 28 treated with any oral, inhaled, or IV antibiotics regardless of potential activity against MRSA | Period ranging from start of Baseline and continuing through Day 28
  Pulmonary exacerbation is defined as having 1 of the major criteria or 2 of the minor signs/symptoms and fulfillment of symptom duration.
  Major criteria:
  1. Absolute decrease in FEV1 of ≥ 10% from Visit 1 (Baseline), unresponsive to albuterol (in participants able to reproducibly perform spirometry)
  2. Oxygen saturation <90% on room air or absolute decrease of ≥ 5% from Visit 1
  3. New lobar infiltrate(s) or atelectasis on chest radiograph
  4. Hemoptysis (more than streaks on more than one occasion in past week)
  Minor signs/symptoms:
  1. Increased work of breathing or respiratory rate
  2. New or increased adventitial sounds on lung exam
  3. Weight loss ≥5% of body weight or decrease across 1 major percentile in weight percentile for age in past 6 months
  4. Increased cough
  5. Decreased exercise tolerance or level of activity
  6. Increased chest congestion or change in sputum
  Signs/symptoms duration: initial symptom must have occurred for at least 5 days.
Proportion of subjects treated with oral, inhaled, and IV antibiotics over the six-month study | Period ranging from start of Baseline and continuing through Month 6
Time to protocol-defined pulmonary exacerbation over the six-month study | Period ranging from start of Baseline and continuing through Month 6
  Pulmonary exacerbation is defined as having 1 of the major criteria or 2 of the minor signs/symptoms and fulfillment of symptom duration.
  Major criteria:
  1. Absolute decrease in FEV1 of ≥ 10% from Visit 1 (Baseline), unresponsive to albuterol (in participants able to reproducibly perform spirometry)
  2. Oxygen saturation <90% on room air or absolute decrease of ≥ 5% from Visit 1
  3. New lobar infiltrate(s) or atelectasis on chest radiograph
  4. Hemoptysis (more than streaks on more than one occasion in past week)
  Minor signs/symptoms:
  1. Increased work of breathing or respiratory rate
  2. New or increased adventitial sounds on lung exam
  3. Weight loss ≥5% of body weight or decrease across 1 major percentile in weight percentile for age in past 6 months
  4. Increased cough
  5. Decreased exercise tolerance or level of activity
  6. Increased chest congestion or change in sputum
  Signs/symptoms duration: initial symptom must have occurred for at least 5 days.
Number of protocol-defined pulmonary exacerbations over the six-month study | Period ranging from start of Baseline and continuing through Month 6
  Pulmonary exacerbation is defined as having 1 of the major criteria or 2 of the minor signs/symptoms and fulfillment of symptom duration.
  Major criteria:
  1. Absolute decrease in FEV1 of ≥ 10% from Visit 1 (Baseline), unresponsive to albuterol (in participants able to reproducibly perform spirometry)
  2. Oxygen saturation <90% on room air or absolute decrease of ≥ 5% from Visit 1
  3. New lobar infiltrate(s) or atelectasis on chest radiograph
  4. Hemoptysis (more than streaks on more than one occasion in past week)
  Minor signs/symptoms:
  1. Increased work of breathing or respiratory rate
  2. New or increased adventitial sounds on lung exam
  3. Weight loss ≥5% of body weight or decrease across 1 major percentile in weight percentile for age in past 6 months
  4. Increased cough
  5. Decreased exercise tolerance or level of activity
  6. Increased chest congestion or change in sputum
  Signs/symptoms duration: initial symptom must have occurred for at least 5 days.
MRSA Culture Status | Day 56
  Proportion of subjects with a negative culture for MRSA at Day 56
Proportion of subjects with >80% compliance for study drug during the first 28 days | Day 28
  Compliance refers to the amount of prescribed medication consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Muhlebach, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (9):
- United States (9):
  - National Jewish Health, Denver, Colorado
  - Indiana University, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - N.C. Memorial Hospital and N.C. Children's Hospital, Chapel Hill, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - University of Washington Medical Center and Seattle Children's, Seattle, Washington

REFERENCES:
- [Background] Muhlebach MS, Beckett V, Popowitch E, Miller MB, Baines A, Mayer-Hamblett N, Zemanick ET, Hoover WC, VanDalfsen JM, Campbell P, Goss CH; STAR-too study team. Microbiological efficacy of early MRSA treatment in cystic fibrosis in a randomised controlled trial. Thorax. 2017 Apr;72(4):318-326. doi: 10.1136/thoraxjnl-2016-208949. Epub 2016 Nov 15. PMID 27852955